CLINICAL TRIAL: NCT07082816
Title: A Phase III, Prospective, Double-Masked, Randomized, Multi-Center, Active-Controlled, Parallel Group Comparison Study Assessing the Ocular Hypotensive Efficacy of Reformulated PG324 Ophthalmic Solution in Subjects With Elevated Intraocular Pressure
Brief Title: Reformulated PG324 Ophthalmic Solution for Intraocular Pressure Reduction
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLR749-C001
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: Glaucoma; OAG; OHT
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — netarsudil; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reformulated PG324 (Experimental): One drop of netarsudil 0.01%/latanoprost 0.005% ophthalmic solution in each eye in the evening for three months
  Interventions: Drug: Netarsudil 0.01%/latanoprost 0.005% ophthalmic solution
- PG324 (Active Comparator): One drop of netarsudil 0.02%/latanoprost 0.005% ophthalmic solution in each eye in the evening for three months
  Interventions: Drug: Netarsudil 0.02%/latanoprost 0.005% ophthalmic solution

INTERVENTIONS:
Drug: Netarsudil 0.01%/latanoprost 0.005% ophthalmic solution — Investigational ophthalmic solution
  Other Names: Reformulated PG324
  Arms: Reformulated PG324
Drug: Netarsudil 0.02%/latanoprost 0.005% ophthalmic solution — Commercially available ophthalmic solution
  Other Names: PG324; Rocklatan®
  Arms: PG324

SUMMARY:
This study is designed to see how safe and effective a new eye drop, called Reformulated PG324, is for lowering eye pressure in people with open-angle glaucoma (OAG) or ocular hypertension (OHT).

DETAILED DESCRIPTION:
About 470 adults with OAG or OHT will be randomly divided into 2 groups. One group will use the new Reformulated PG324 eye drops, and the other group will use the marketed PG324 eye drops. This study will be double-masked, so neither the researcher nor the participant will know which eye drop was administered. The expected individual duration of participation is approximately 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes;
* Unmedicated intraocular pressure measurements in the study eye as specified in the protocol;
* Corrected distance visual acuity equal to or better than 20/100 in the study eye.

Key Exclusion Criteria:

* Current use of more than 2 ocular hypotensive medications within 30 days;
* Intraocular pressure greater than 36 millimeters mercury (mmHg) at Screening;
* Use of topical ocular medication of any kind within 5 days of Screening or throughout the study with the exception of ocular hypotensive medications (must be washed out).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Intraocular Pressure at each timepoint post-randomization | Week 2, Week 6, Month 3 at 08:00, 10:00, 16:00 hours
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer and recorded in millimeters mercury (mmHg). IOP will be calculated as the mean of two readings or the median of three readings at each timepoint.

SECONDARY OUTCOMES:
Proportion of subjects with moderate to severe conjunctival hyperemia as assessed by biomicroscopy | Up to Month 3/study exit
  The subject will undergo a slit lamp examination at all visits, except for dispensing visits. The presence of moderate to severe conjunctival hyperemia (redness) will be recorded.
Proportion of subjects with conjunctival hyperemia adverse events | Up to Month 3/study exit
  Occurrences of conjunctival hyperemia (redness) adverse events, either subject or investigator reported, will be recorded at each visit.
Mean change from diurnally adjusted baseline IOP at each timepoint post-randomization | Baseline (Day 1), Week 2, Week 6, Month 3 at 08:00, 10:00, 16:00 hours
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer and recorded in millimeters mercury (mmHg). IOP will be calculated as the mean of two readings or the median of three readings at each timepoint. Change is defined as the follow-up (Week 2, Week 6, and Month 3) minus baseline (Day 1) at each timepoint.
Percent change from diurnally adjusted baseline IOP at each timepoint post-randomization | Baseline (Day 1), Week 2, Week 6, Month 3 at 08:00, 10:00, 16:00 hours
  Intraocular pressure (IOP) will be measured with a Goldmann tonometer and recorded in millimeters mercury (mmHg). IOP will be calculated as the mean of two readings or the median of three readings at each timepoint. Change is defined as the follow-up (Week 2, Week 6, and Month 3) minus baseline (Day 1) at each timepoint.
Mean TSS-IOP scores at Month 3 | Month 3
  The Treatment Satisfaction Survey for Intraocular Pressure (TSS-IOP) module is a 15-item questionnaire designed to assess subject satisfaction with ocular hypotensive medication(s). Subjects will respond to each item using a 5-, 6-, or 7-point Likert Scale. Individual scores will be computed by adding the scale values of items within a satisfaction category and transforming the resulting value into a score between 0 and 100. Higher scores are indicative of greater satisfaction. The questionnaire will be self-administered.
Mean Changes in TSS-IOP scores from Screening to Month 3 | Month 3
  The Treatment Satisfaction Survey for Intraocular Pressure (TSS-IOP) module is a 15-item questionnaire designed to assess subject satisfaction with ocular hypotensive medication(s). Subjects will respond to each item using a 5-, 6-, or 7-point Likert Scale. Individual scores will be computed by adding the scale values of items within a satisfaction category and transforming the resulting value into a score between 0 and 100. Higher scores are indicative of greater satisfaction. The questionnaire will be self-administered.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (30):
- United States (30):
  - Trinity Research Group, Dothan, Alabama
  - Eye Doctors of Arizona, Phoenix, Arizona
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - United Medical Research Institute, Inglewood, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Sacramento Eye Consultants, Sacramento, California
  - Central Florida Eye Specialists, DeLand, Florida
  - Glaucoma Specialists of South Florida, Delray Beach, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Central Florida Eye Associates, Lakeland, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - Lee Shettle Eye, Largo, Florida
  - North Georgia Eye Associates, Gainesville, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - NorthEast Eye Research Associates, LLC, Westborough, Massachusetts
  - Coldwater Vision Research, Coldwater, Mississippi
  - Las Vegas Eye Institute, Henderson, Nevada
  - Rochester Ophthalmological Group, Rochester, New York
  - Albemarle Eye Center, Elizabeth City, North Carolina
  - Oculus Research, Inc., Garner, North Carolina
  - CORE, Inc., Shelby, North Carolina
  - Midwest Eye Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No